CLINICAL TRIAL: NCT01775852
Title: Brief, Behavioral Intervention of ACT & Illness Management for Comorbid Migraine and Depression
Brief Title: Brief Behavioral Intervention for Comorbid Migraine and Depression
Acronym: ACT-IM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lilian N. Dindo (Other)
Responsible Party: Sponsor-Investigator, Lilian N. Dindo, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201004763; ICTS-01 (Other Grant/Funding Number: University of Iowa, ICTS)
Record Dates: First submitted 2012-01-09; First posted 2013-01-25 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Migraine; Depression
Keywords: Acceptance and Commitment Therapy (ACT); Depression; Illness Management; Behavioral treatment; Impairment
MeSH Terms: conditions — Migraine Disorders; Depression | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT-IM (Active Comparator): The ACT-IM arm is a brief, one-day intervention that includes two components: 1) Illness Management for Migraine and, 2) Acceptance and Commitment Therapy for emotional difficulties that go along with, or are exacerbated by migraine.
  Interventions: Behavioral: ACT-IM
- Waitlist/Treatment as Usual (No Intervention): The Waitlist/Treatment as Usual (WL/TAU)condition completes the same assessments as the active treatment group but does not undergo the active treatment (workshop) until after the 12-week follow-up visit. At that point, the WL/TAU participants are given the opportunity to join a treatment workshop.

INTERVENTIONS:
Behavioral: ACT-IM — 1 hour discussion about migraine management (IM) and 5 hours of group therapy based on Acceptance and Commitment Therapy (ACT). IM covers symptoms and triggers for worsening of migraine symptoms, how to use migraine medications, medication overuse headache, etc. The ACT intervention includes: 1) Behavioral Change Training and; 2) Mindfulness and Acceptance Training emphasizing new ways of managing troubling thoughts, feelings, and physical sensations.
  Other Names: Acceptance and Commitment Therapy; Illness Management
  Arms: ACT-IM

SUMMARY:
The purpose of this research study is to examine whether a one-day group workshop, integrating principles from Acceptance and Commitment Therapy with Migraine Education, will result in improvements in depressive symptoms and functioning impairment in patients with comorbid migraine and depression.

DETAILED DESCRIPTION:
Migraine affects approximately 35 million US residents (Bigal & Lipton, 2009) and is associated with excruciating headache and marked functional impairment. Epidemiological and clinical research has shown that people with migraine suffer from psychiatric disorders at a disproportionately higher rate than individuals without. Depression, in particular, is 3-5 times more common in migraine patients than in non-migraineurs. The comorbidity of depression and migraine is a major health concern as it results in poorer prognosis, remission rate, and response to treatment. In addition, an increase in the severity of migraine is associated with a parallel rise in the severity and treatment resistance of comorbid depression.

Recent research in behavioral medicine suggests that the pain experience per se does not necessarily lead to depression or impairment. Instead, it is the preoccupation with avoiding aversive stimuli associated with pain (i.e., activities, places, movements) that results in depression and disability (e.g., McCracken et al., 2005). Therefore, given that patients with migraine and/or depression exhibit more avoidance behaviors and lower activity levels than healthy controls (e.g., Stronks et al., 2004), an intervention aimed at optimizing willingness and acceptance and minimizing behavioral avoidance may be beneficial at improving both their depression and migraine and, consequently, their daily functioning.

Acceptance and Commitment Therapy (ACT) is an empirically based behavioral therapy that incorporates acceptance and mindfulness strategies with behavioral change strategies. ACT (in group and in individual settings) is effective in treating psychiatric disorders commonly associated with migraine, including depression, anxiety, and stress (e.g., Hayes, 2001) as well as chronic illnesses like pain and diabetes (Dahl et al, 2004; Gregg et al., 2006). Importantly, ACT resulted in positive long-term outcomes even when presented in brief form. For example, a two-day ACT workshop, in a group setting, led to improvements in depression and distress experienced by parents of children diagnosed with autism and these gains were retained 3 months later. Parents also exhibited a reduction in avoidance behaviors (Blackledge & Hayes, 2006).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* 4 to 12 migraines in the previous month
* Major or Minor Depression
* English-speaking

Exclusion Criteria:

* Patients with other major psychiatric disorders such as bipolor disorder, schizophrenia, and current illicit drug use.
* Patients with major head injuries.
* Patients with serious medical illnesses.
* Patients who have started a new medication in previous 4 weeks or plan on starting a new medication in the next 4 weeks.
* Patients expressing significant suicidal ideation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Dindo, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] Bigal ME, Lipton RB. The epidemiology, burden, and comorbidities of migraine. Neurol Clin. 2009 May;27(2):321-34. doi: 10.1016/j.ncl.2008.11.011. PMID 19289218
- [Background] Breslau N, Lipton RB, Stewart WF, Schultz LR, Welch KM. Comorbidity of migraine and depression: investigating potential etiology and prognosis. Neurology. 2003 Apr 22;60(8):1308-12. doi: 10.1212/01.wnl.0000058907.41080.54. PMID 12707434
- [Background] Blackledge, J.T. & Hayes, S.C. Using Acceptance and Commitment Training in the support of parents of children diagnosed with Autism. Child and Family Behavior Therapy. 2006;28(1):1-18.
- [Background] Dahl, J., Wilson, K.G., Nilsson, A. Acceptance and Commitment Therapy and the treatment of persons at risk for long-term disability resulting from stress and pain symptoms: A preliminary randomized trial. Behavior Therapy. 2004;35:785-801.
- [Background] Gregg JA, Callaghan GM, Hayes SC, Glenn-Lawson JL. Improving diabetes self-management through acceptance, mindfulness, and values: a randomized controlled trial. J Consult Clin Psychol. 2007 Apr;75(2):336-43. doi: 10.1037/0022-006X.75.2.336. PMID 17469891
- [Background] Hayes SC. Acceptance and Commitment Therapy, Relational Frame Theory, and the Third Wave of Behavioral and Cognitive Therapies - Republished Article. Behav Ther. 2016 Nov;47(6):869-885. doi: 10.1016/j.beth.2016.11.006. Epub 2016 Nov 10. PMID 27993338
- [Background] Lake AE 3rd, Rains JC, Penzien DB, Lipchik GL. Headache and psychiatric comorbidity: historical context, clinical implications, and research relevance. Headache. 2005 May;45(5):493-506. doi: 10.1111/j.1526-4610.2005.05101.x. PMID 15953266
- [Background] Lundgren T, Dahl J, Melin L, Kies B. Evaluation of acceptance and commitment therapy for drug refractory epilepsy: a randomized controlled trial in South Africa--a pilot study. Epilepsia. 2006 Dec;47(12):2173-9. doi: 10.1111/j.1528-1167.2006.00892.x. PMID 17201719
- [Background] McCracken LM, Vowles KE, Eccleston C. Acceptance-based treatment for persons with complex, long standing chronic pain: a preliminary analysis of treatment outcome in comparison to a waiting phase. Behav Res Ther. 2005 Oct;43(10):1335-46. doi: 10.1016/j.brat.2004.10.003. Epub 2005 Jan 7. PMID 16086984
- [Background] Stronks DL, Tulen JH, Bussmann JB, Mulder LJ, Passchier J. Interictal daily functioning in migraine. Cephalalgia. 2004 Apr;24(4):271-9. doi: 10.1111/j.1468-2982.2004.00661.x. PMID 15030535
- See also: Online, screening survey. — http://goo.gl/FFged
- See also: University of Iowa Hospitals & Clinics — http://uihealthcare.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACT-IM | Waitlist/Treatment as Usual
Started | 31 | 14
Completed | 31 | 13
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACT-IM | Waitlist/Treatment as Usual | Total
Number analyzed (Participants) | 31 | 14 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (13.3) | 33.5 (12.9) | 33 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 12 | 42
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hamilton Depression Rating Scale (HAM-D) From Baseline to 12 Week Follow-up
Description: The HAM-D is a structured clinical interview for assessing depression severity. Outcome measure will be change from Baseline in Hamilton Depression Rating Scale at 12 week (3 month) follow-up from baseline.
  Measure is scored by adding individual items and attaining an overall severity score. Scores range from 0 to 53, with higher values signifying a higher level of depression severity (and thus a worse outcome). A score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial.
Time Frame: 12 week change from baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT-IM | Waitlist/Treatment as Usual
Number analyzed (Participants) | 31 | 14
units on a scale | -15.1 (1.6) | -4.3 (2.5)

2. Secondary Outcome: Mean Change Score in HDI (Headache Disability Inventory) From Baseline to 12 Weeks.
Description: The HDI is useful in assessing the impact of headache, and its treatment, on daily living. 25 self-report items are rated with answers as "Yes" (4 points), "Sometimes" (2 Points), and "No" (0 points). All items are then added together to create an overall score which can range from 0 (no impact), to 100 (severe impact) of headache on daily life.
  A 29 point change (95% confidence interval) or greater in the total score from test to retest must occur before the change can be attributed to treatment effects.
Time Frame: 12 week change from baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT-IM | Waitlist/Treatment as Usual
Number analyzed (Participants) | 31 | 14
units on a scale | -27.9 (3.4) | -10.7 (5.2)

3. Secondary Outcome: Mean Change on Short Form Health Survey (SF-36) From Baseline to 12 Week Follow-up.
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Change at 12 week follow-up from baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT-IM | Waitlist/Treatment as Usual
Number analyzed (Participants) | 31 | 14
units on a scale | 17.0 (2.5) | 7.7 (3.8)

4. Secondary Outcome: Mean Change of World Health Organization Disability Assessment (WHO-DAS) From Baseline to 12-week Follow up.
Description: The WHODAS contains 36 items on functioning and disability with a recall period of 30 days covering 7 domains: Understanding and Communicating (6 items), Getting around (5 items), Self-care (4 items), Getting along with others (5 items), Life activities: household (4 items), Life activities: work/school (4 items), and Participation in society (8 items). Response options go from 1 (no difficulty) to 5 (extreme difficulty or can not do).
  WHODAS domain scores are computed for each domain by adding the item responses together. A global score is then computed by summing all domains together, and transforming them into a range from 0 to 100, with higher scores indicating higher levels of disability (0= no disability, 100= full disability).
Time Frame: Change at 12 week follow-up from baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ACT-IM | Waitlist/Treatment as Usual
Number analyzed (Participants) | 31 | 14
units on a scale | -9.1 (2) | -.3 (2.9)

ADVERSE EVENTS:
Arm/Group | ACT-IM | Waitlist/Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/14
Other Adverse Events (participants affected / at risk) | 0/31 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No